CLINICAL TRIAL: NCT03992183
Title: TH-146: Cancer Associated Macrophage-Like (CAML) Cells to Enhance Detection of Early Stage Lung Cancer
Brief Title: Utility of CAML as Diagnostic for Early Stage Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Creatv Microtech, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: TH-146
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Nodule, Multiple; Pulmonary Nodule, Solitary
Keywords: CAML; Early Detection
MeSH Terms: conditions — Multiple Pulmonary Nodules; Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two 10cc of blood per draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary Objective Determine the prevalence of CAMLS in patients with pulmonary nodules.

Secondary Objectives Determine the positive and negative predictive value of CAMLS in patients with pulmonary nodules who undergo biopsy.

Model combinations of clinical factors with the presence/absence of CAMLS to refine strategies for assessment of patients with pulmonary nodules. Evaluate whether these measures result in enhanced T-cell activity and/or NK cell function and number

ELIGIBILITY:
Inclusion Criteria:

* Referral for a pulmonary nodule that has not yet been biopsied and that meets the definition of an "indeterminate" nodules (i.e. 0.8-3.0 cm).
* No prior diagnosis of lung cancer or other invasive malignancy within the past 5 years.
* No history of rheumatologic disease.
* Age > 18 years.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

* Patients with active, known or suspected autoimmune disease.
* Prior diagnosis of lung cancer or other invasive malignancy within the past 5 years.
* Uncontrolled intercurrent illness that would increase the risk of toxicity or limit compliance with study requirements. This includes but is not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV-positive patients on combination antiretroviral therapy are ineligible because of the abnormal immune response that results from HIV disease (testing is not required).
* Patients should be excluded if they are known to be positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection (testing is not required).
* Subjects with any history of interstitial lung disease or a history of > or = to grade 2 radiation pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be drawn from pulmonary nodule clinics at the Fox Chase Cancer Center and the VAMC Philadelphia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Determination of prevalence pf CAMLs in Pulmonary modules | During the first 2 years of study
  Laboratory studies performed on blood drawn at Creatv Microtech will determine the prevalence of CAMLS in pulmonary nodules.

SECONDARY OUTCOMES:
Determination of positive and negative predictive value, sensitivity and specificity of CAMLS in patients with pulmonary nodules who undergo biopsy | Through study completion, an average of 3 years
  Positive Predictive Value and Negative Predictive Value, sensitivity and specificity at the initial screen will be computed for the entire study population.
Model combinations of clinical factors with the presence/absence of CAMLs to refine strategies for assessment of patients with pulmonary nodules. Evaluate whether measures result in enhanced T-cell activity/Natural Killer (NK) cell function and number | Through study completion, a maximum of 3 years
  Bidimensional measurements of lung nodules done by a radiologist or pulmonary physician from CT scans with 5mm (or less) cuts, using lung windows in the axial plane

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT03992183/Prot_SAP_000.pdf